CLINICAL TRIAL: NCT00675207
Title: Comparison of Brimonidine 0.15% Purite, Dorzolamide 2%, and Brinzolamide 1% as Adjunctive Therapy to Prostaglandin Analogs
Brief Title: Comparison of Brimonidine Purite, Dorzolamide, and Brinzolamide as Adjunctive Therapy to Prostaglandin Analogs
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Northwestern Ophthalmic Institute S.C. (Other)
Collaborators: Research to Prevent Blindness (Other)
Responsible Party: Thomas E. Bournias, Northwestern Ophthalmic Institute S.C.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NWOIADJ 2006
Record Dates: First submitted 2008-05-06; First posted 2008-05-08 (Estimated); Last update posted 2008-05-08 (Estimated); Status verified 2008-05

CONDITIONS: Primary Open Angle Glaucoma; Ocular Hypertension
Keywords: glaucoma; ocular hypertension; adjunctive treatment; prostaglandin; prostaglandin analog; brimonidine; dorzolamide; brinzolamide; alpha agonist; carbonic anhydrase inhibitor; intraocular pressure
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension; Glaucoma | interventions — dorzolamide; brinzolamide

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator): Brimonidine purite 0.15%
  Interventions: Drug: Brimonidine purite 0.15%
- 2 (Active Comparator): Dorzolamide 2%
  Interventions: Drug: Dorzolamide 2%
- 3 (Active Comparator): Brinzolamide 1%
  Interventions: Drug: Brinzolamide 1%

INTERVENTIONS:
Drug: Brimonidine purite 0.15% — A single drop of brimonidine purite 0.15% ophthalmic solution administered topically in the eye 3 times daily.
  Other Names: Alphagan P 0.15%
  Arms: 1
Drug: Dorzolamide 2% — A single drop of dorzolamide 2% ophthalmic solution administered topically in the eye 3 times daily.
  Other Names: Trusopt
  Arms: 2
Drug: Brinzolamide 1% — A single drop of brinzolamide 1% ophthalmic solution administered topically in the eye 3 times daily.
  Other Names: Azopt
  Arms: 3

SUMMARY:
The purpose of this study is to compare the efficacy of brimonidine Purite, dorzolamide, and brinzolamide in reducing intraocular pressure when added to prostaglandin analog therapy (bimatoprost, latanoprost, or travoprost) in patients with glaucoma or ocular hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary open-angle glaucoma or ocular hypertension.
* Must be over 40 years of age.
* Intraocular pressure must be 18 mm Hg or higher after 6 weeks of treatment (run-in) with a prostaglandin analog (bimatoprost, latanoprost, or travoprost).

Exclusion Criteria:

* History of angle closure or narrow angle.
* Previous intraocular surgery.
* Laser trabeculoplasty within 3 months prior to screening.
* History of uveitis or intraocular inflammation.
* Use of medications other than the study medications that are known to affect IOP (e.g., beta-blockers, steroids, or angiotensin II blockers) within 3 months of study entry or during the study.
* Intolerance of or hypersensitivity to prostaglandin analogs, sulfonamides, alpha-agonists, or the preservative benzalkonium chloride.
* Women of childbearing age who are pregnant or not using contraception.

Min Age: 41 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2006-01; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Intraocular pressure | Measurements at peak and trough effect (10 am and 4 pm) at baseline, month 1, and month 4

CONTACTS AND LOCATIONS:
Overall Officials: Thomas E. Bournias, MD, Principal Investigator — Northwestern Ophthalmic Institute S.C.
Locations (1):
- Northwestern Ophthalmic Institute S.C., Glenview, Illinois, United States